CLINICAL TRIAL: NCT03728842
Title: Blood Drawing for Study of Peripheral Blood T-lymphocytes and Other Parameters in Patients With Metastatic Melanoma and Renal Cell Cancer With Spontaneous Regression
Brief Title: Spontaneous Regression in Metastatic Melanoma and Renal Cell Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Theodore Logan, Associate Professor of Medicine, Indiana University School of Medicine
Other Study IDs: IUCRO-0042; 1011003667 (Other: Indiana University IRB)
Record Dates: First submitted 2018-10-05; First posted 2018-11-02 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Melanoma; Renal Cell Carcinoma
Keywords: metastatic disease; spontaneous regression
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Neoplasm Metastasis; Remission, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spontaneous regression: Patients must have metastatic melanoma or renal cell cancer with spontaneous regression.
  Interventions: Other: Blood collection for laboratory studies; Other: Data collection from medical record

INTERVENTIONS:
Other: Blood collection for laboratory studies — Peripheral whole blood will be collected
Other: Data collection from medical record — Clinical data such as demographics and cancer characteristics, history and treatment will be collected

SUMMARY:
The purpose of this study is to collect blood and clinical data from patients with metastatic melanoma and renal cell cancer who have experienced spontaneous regression for studies of immune response and other factors that may influence these occurrences.

DETAILED DESCRIPTION:
Spontaneous regression in patients with metastatic cancer is an incredibly rare event. It has been described after infection in cancer patients and also rarely in patients with renal cell cancer (usually after resection of the renal primary) and, less commonly, in patients with metastatic melanoma.

Primary Objective To collect peripheral blood from patients with metastatic melanoma and renal cell cancer and spontaneous regression for studies of immune response and other studies.

Secondary Objective To collect clinical data from subjects registered to this study. Clinical data collection will include demographics and cancer characteristics, history and treatment.

ELIGIBILITY:
Inclusion Criteria

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Patients must have metastatic melanoma or renal cell cancer with spontaneous regression.
4. Willingness to undergo phlebotomy for research blood samples

Exclusion Criteria

1. Concurrent disease or condition that would make the patient inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety
2. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic melanoma and renal cell cancer and spontaneous regression.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2004-01-04 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of blood samples collected | 1 year
  samples collected from metastatic melanoma and renal cell cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Logan, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided